CLINICAL TRIAL: NCT03016728
Title: Exploring the Feasibility, Safety, and Potential Benefits of a 12-week Home-based Physical Activity Intervention
Brief Title: Physical Activity for Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, PhD, Assistant Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ottawa
Record Dates: First submitted 2016-12-24; First posted 2017-01-11 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Adolescent and Young Adult Cancer Survivors
Keywords: exercise; physical activity; pilot study; randomized controlled trial; cancer; adolescent and young adult; AYA
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): Participants in the experimental arm (i.e., physical activity) will be asked to complete the 12-week home-based physical activity program and to complete all study assessments.
  Interventions: Behavioral: Physical Activity
- Wait-List Control (No Intervention): Participants in the no intervention arm (i.e., wait-list control) will be asked to maintain their usual lifestyle activities and to complete all study assessments. Participants in this arm will be provided with the 12-week home-based physical activity program in the exact same way as participants in the experimental arm (i.e., physical activity) at the end of the study.

INTERVENTIONS:
Behavioral: Physical Activity — Participants will receive a 12-week home-based physical activity program that has been individualized using their baseline assessment results. The program will be comprised of aerobic training (2 days/week) and resistance training (2 days/week). The aerobic training will be performed unsupervised. The resistance training will be performed under the supervision of a study team member (who will visit participants homes) for the first 6 weeks to ensure proper form and safety.
  Arms: Physical Activity

SUMMARY:
More adolescents and young adults are surviving cancer than ever before. Many endure negative effects related to their cancer and its treatment, which reduces their quality of life and functioning. Physical activity is one strategy that has been shown to promote quality of life amongst cancer survivors. However, very little research has focused on adolescent and young adult cancer survivors. Therefore, the purpose of this pilot randomized controlled trial is to explore the feasibility, safety, and potential benefits of a 12-week home-based physical activity intervention in adolescent and young adult cancer survivors.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Have been diagnosed with cancer for the first time between the ages of 15 and 39 years;
2. Have completed cancer treatment within 5 years;
3. Currently between the ages of 15 to 44 years;
4. Have no current evidence of progressive disease, secondary cancer (i.e., cancer cells that have spread from the primary cancer), or second cancers (i.e., a new different cancer);
5. Live within 100 km of the University of Ottawa;
6. Be inactive or insufficiently active as determined by a single item screening question (i.e., participants must respond "no" to the following question: are you currently engaging in moderate physical activity, defined as activity that increases your heart rate and causes you to sweat, on 3 or more days a week?). Screening participants based on their level of physical activity will ensure only those individuals for whom the intervention will have the largest effect are recruited;
7. Able to read, understand, and provide informed consent in English;
8. Ready for physical activity as indicated by answering Physical Activity Readiness Questions (PAR-Q). If participants are not ready for physical activity as determined by the PAR-Q they will need to complete a Physical Activity Readiness Medical Examination Form.

EXCLUSION CRITERIA:

1. Physical impairments precluding participation in physical activity;
2. Unwilling or unable to sign the Participant Informed Consent Form;
3. Received a diagnosis of brain cancer or thyroid cancer. Brain cancer survivors will be excluded as a function of the cognitive impairments associated with their diagnosis and treatment and thyroid cancer survivors will be excluded due to the vastly different treatment regimens. That is, both of these cancers may result in different physical, psychological/emotional, and social effects that could impact the outcomes of interest.

Eligible participants who want to participate in the other pre-specified outcome measures to assess cognitive functioning must also meet the following additional inclusion/exclusion criteria.

ADDITIONAL INCLUSION CRITERIA:

1. Right-handedness, because language is lateralized and has been shown to be left side dominant (for right handers) during fMRI tasks;
2. Able to read, understand, and provide informed consent in English for the additional assessments.

ADDITIONAL EXCLUSION CRITERIA:

1. Metal implants (e.g., pacemaker) or metal dental work (aside from fillings) that would preclude scanning;
2. Claustrophobia;
3. Poor eyesight (not correctable with contact lenses) that precludes viewing stimuli presented in the scanner;
4. Lower back pain that would preclude a person from lying relatively still for one hour;
5. Substance use disorder as assessed by a single item question (i.e., participants must respond "no" to the following question: Have you been told, in the last five years, by your healthcare provider that you have a substance use disorder?).

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Recruitment Rates | Through study completion, an average of 12-24 weeks
  The number of eligible participants who enrol in the study out of the number who are referred.
Retention Rates | Through study completion, an average of 12-24 weeks
  The number of participants completing the intervention and all scheduled assessments.
Adherence Rates | Through study completion, an average of 12-24 weeks
  The number of physical activity sessions engaged in out of the total recommended as part of the intervention.
Number of Participants with Adverse Events | Through study completion, an average of 12-24 weeks
  The number of participants reporting or presenting adverse events (e.g., injury) that occurs as a result of participating in the physical activity intervention and/or its assessments.

SECONDARY OUTCOMES:
Physical Activity Behaviour: Daily Physical Activity Logbook | Through study completion, an average of 12-24 weeks
  Change in daily self-reported daily physical activity from baseline, to mid-intervention, to post-intervention, to follow-up (if applicable; i.e., if participant consents and is eligible to participate in the additional assessments testing cognitive functioning).
Physical Activity Behaviour: Leisure Time Exercise Questionnaire (Godin & Shephard, 1985) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12), follow-up (week 24)
  Change in self-reported physical activity (over the past 7 days) from baseline, to mid-intervention, to post-intervention, to follow-up (if applicable; i.e., if participant consents and is eligible to participate in the additional assessments testing cognitive functioning).
Physical Activity Behaviour: 7-Day Accelerometer Wear (Objective Physical Activity Behaviour) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12), follow-up (week 24)
  Change in objective levels of physical activity as measured by accelerometers (Actigraph wGT3XP-BT), which will be worn for a 7 day period from baseline, to mid-intervention, to post-intervention, to follow-up (if applicable; i.e., if participant consents and is eligible to participate in the additional assessments testing cognitive functioning).
Resting Heart Rate | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in resting heart rate, as measured by a heart rate monitor (Polar A300), from baseline, to mid-intervention, to post-intervention.
Blood Pressure | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in resting blood pressure, using a blood pressure monitor (HealthSmart Digital Blood Pressure Monitor), from baseline, to mid-intervention, to post-intervention.
Body Composition: Body Mass Index | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in body mass as determined by a Tanita scale (TBF-310 GS) that uses bioelectrical impedance to assess body composition from baseline, to mid-intervention, to post-intervention.
Aerobic Capacity: 6-Minute Walk Test (CSEP, 2013; Irwin, 2012) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in aerobic capacity (i.e., total distance walked in 6 minutes) from baseline, to mid-intervention, to post-intervention.
Musculoskeletal Strength: Combined Grip Strength using a Handheld Dynamometer (CSEP, 2013; Irwin, 2012) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in musculoskeletal strength (i.e., force exerted in kilograms on the handheld dynamometer) from baseline, to mid-intervention, to post-intervention.
Muscular Endurance: 30-Second Sit to Stand Test (Rikli & Jones, 2001) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in muscular endurance (i.e., number of times participants can stand from a seated position in 30 seconds) from baseline, to mid-intervention, to post-intervention.
Self-Efficacy: Single-Item Version of the Exercise Self-Efficacy Scale (McAuley, 1993) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in participants self-reported self-efficacy from baseline, to mid-intervention, to post-intervention.
Physical Competence and Physical Self-Esteem: Physical Self-Description Questionnaire Short-Form Appearance, Strength, Endurance, Body Fat, and Physical Self-Esteem scales (Marsh, Martin, & Jackson, 2010) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in participants self-reported physical competence and physical self-esteem from baseline, to mid-intervention, to post-intervention.
Global Self-Esteem: Rosenberg Global Self-Esteem Scale (Rosenberg, 1965) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in participants self-reported global self-esteem from baseline, to mid-intervention, to post-intervention.
Body Image: Multidimensional Body-Self Relations Questionnaire Appearance Evaluation and Body Areas Satisfaction scales (Cash, 2000) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in participants self-reported body image from baseline, to mid-intervention, to post-intervention.
Posttraumatic Growth: Posttraumatic Growth Inventory (Tedeschi & Calhoun, 1996) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in participants self-reported posttraumatic growth from baseline, to mid-intervention, to post-intervention.
Quality of Life: Medical Outcomes Study 36-Item Short-Form Health Survey (Ware & Sherbourne, 1992) | Baseline (week 0), mid-intervention (weeks 6), post-intervention (week 12)
  Change in participants self-reported quality of life from baseline, to mid-intervention, to post-intervention.
Participants Experiences: Qualitative Interviews | Baseline (week 0), post-intervention (week 12)
  Participants experiences in the intervention (i.e., with physical activity if in the experimental arm or with engaging in their usual lifestyle if in the wait-list control arm) and subsequent changes, if any, in behavioural, physical, psychological, and quality of life outcomes as explored via qualitative interviews (following an interview schedule containing a series of open-ended questions and probes) from baseline to post-intervention.

OTHER OUTCOMES:
Cognitive Functioning: Single Open-Ended Question | Baseline (week 0), post-intervention (week 12), follow-up (week 24)
  Change in participants responses to a single open-ended question: "Do you ever feel like you have a hard time thinking and/or remembering?" from baseline, to post-intervention, to follow-up.
  NOTE: Once recruited to the main trial, participants will have the option to participate in additional assessments testing cognitive functioning. If interested, participants must meet additional inclusion/exclusion criteria for the additional assessments.
Cognitive Functioning: Magnetic Resonance Imaging (MRI) Scans | Baseline (week 0), post-intervention (week 12), follow-up (week 24)
  Change in participants cognitive functioning, as assessed by a structural scan, a resting state functional MRI (fMRI) procedure, four fMRI tasks, and a diffusion tensor imaging sequence (lasting approximately 60 minutes), from baseline, to post-intervention, to follow-up.
  NOTE: Once recruited to the main trial, participants will have the option to participate in additional assessments testing cognitive functioning. If interested, participants must meet additional inclusion/exclusion criteria for the additional assessments.
Socio-Demographic and Medical Information Questionnaire | Baseline (week 0)
  The socio-demographic and medical information collected will be used to describe the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brunet, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Canadian Society for Exercise Physiology (CSEP). CSEP-Physical activity training for health (CSEP-PATH). Ottawa, ON: CSEP, 2013.
- [Background] Irwin, ML. American College of Sports Medicine's guide to exercise and cancer survivorship. Champaign, IL: Human Kinetics, 2012.
- [Background] Rikli R, Jones J. Senior fitness test manual. Champaign, IL: Human Kinetics, 2001.
- [Background] McAuley E. Self-efficacy and the maintenance of exercise participation in older adults. J Behav Med. 1993 Feb;16(1):103-13. doi: 10.1007/BF00844757. PMID 8433355
- [Background] Marsh HW, Martin AJ, Jackson S. Introducing a short version of the physical self description questionnaire: new strategies, short-form evaluative criteria, and applications of factor analyses. J Sport Exerc Psychol. 2010 Aug;32(4):438-82. doi: 10.1123/jsep.32.4.438. PMID 20733208
- [Background] Rosenberg M. Soceity and adolescent self-image. Princeton, NJ: Princeton University Press, 1965.
- [Background] Cash TF. The multidimensional body-self relations questionnaire. MBSRQ Users' Manual 3rd Revision. Available: http://www.body-images.com, 2000.
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Derived] Wurz A, Ayson G, Smith AM, Brunet J. A proof-of-concept sub-study exploring feasibility and preliminary evidence for the role of physical activity on neural activity during executive functioning tasks among young adults after cancer treatment. BMC Neurol. 2021 Aug 4;21(1):300. doi: 10.1186/s12883-021-02280-y. PMID 34344355
- [Derived] Wurz A, Price J, Brunet J. Understanding adolescents' and young adults' self-perceptions after cancer treatment in the context of a two-arm, mixed-methods pilot randomized controlled physical activity trial. Support Care Cancer. 2021 Aug;29(8):4439-4450. doi: 10.1007/s00520-020-05974-0. Epub 2021 Jan 15. PMID 33449169
- [Derived] Wurz A, Brunet J. Exploring the feasibility and acceptability of a mixed-methods pilot randomized controlled trial testing a 12-week physical activity intervention with adolescent and young adult cancer survivors. Pilot Feasibility Stud. 2019 Dec 20;5:154. doi: 10.1186/s40814-019-0530-6. eCollection 2019. PMID 31890266